CLINICAL TRIAL: NCT06042660
Title: Comorbidity Burden and Use of Concomitant Medications at CML Diagnosis: A Retrospective Analysis of 527 Patients From the Polish Adult Leukemia Group Registry
Brief Title: Comorbidity Burden and Use of Concomitant Medications at CML Diagnosis
Status: Completed | Type: Observational
Sponsor: Polish Adult Leukemia Group (Other)
Responsible Party: Principal Investigator, Anna Krec, Project Manager of Polish Adult Leukemia Group, Polish Adult Leukemia Group
Other Study IDs: PALG CML Comorbidity
Record Dates: First submitted 2023-09-11; First posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Chronic Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- newly diagnosed CML patients
  Interventions: Other: the prevalence of comorbid conditions

INTERVENTIONS:
Other: the prevalence of comorbid conditions — analysis of history of comorbidities at the time of CML diagnosis

SUMMARY:
The aim of the retrospective study was to further characterize the prevalence of comorbid conditions as well as the use of concomitant medications in newly diagnosed CML patients in a real-world setting. Hematologists from ten Polish hematological tertiary care centers were asked to analyze medical records for all consecutive CML patients diagnosed with chronic phase CML between January 1st 2005 and December 31st 2014.

DETAILED DESCRIPTION:
All three TKIs used as first line treatment of CML, (imatinib, dasatinib and nilotinib), may be associated with the so called "off-target" effects causing specific adverse events (AEs).

Interestingly, some co-morbidities may predispose towards developing these specific TKIs' "offtarget" AEs.

The aim of the retrospective study was to further characterize the prevalence of comorbid conditions as well as the use of concomitant medications in newly diagnosed CML patients in a real-world setting. Hematologists from ten Polish hematological tertiary care centers were asked to analyze medical records for all consecutive CML patients diagnosed with chronic phase CML between January 1st 2005 and December 31st 2014. Data were collected through on-line case report form of the Polish Adult Leukemia Group (PALG) Registry. Baseline patients' characteristics including sex, age, body mass index (BMI), risk group according to Sokal score, as well as comorbidities and concomitant therapies, were recorded at the time of CML diagnosis. The study was conducted in accordance with the provisions of the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* 1) age ≥ 18 years; 2) diagnosis of chronic phase CML between January 1st 2005 and December 31st 2014.

Exclusion Criteria:

* primary diagnosis of CML in accelerated or blastic phase

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with diagnosis of chronic phase CML diagnosed between January 1st and December 31st 2014, treated with TKI (imatinib, dasatinib, nilotynib)
Sampling Method: Non-Probability Sample
Enrollment: 527 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
the prevalence of comorbid conditions in newly diagnosed CML patients | February - July 2016
  data collected through an on-line questionnaire, descriptive data
the number of concomitant medications in newly diagnosed CML patients | February - July 2016
  data collected through an on-line questionnaire, descriptive data

REFERENCES:
- [Result] Gora-Tybor J, Sacha T, Waclaw J, Niesiobedzka-Krezel J, Grzybowska-Izydorczyk O, Medras E, Deren-Wagemann I, Patkowska E, Seferynska I, Lewandowski K, Wache A, Blajer-Olszewska B, Watek M, Kotwica-Mojzych K, Wasilewska E, Warzocha K, Jamroziak K. Comorbidity Burden and Use of Concomitant Medications at CML Diagnosis: A Retrospective Analysis of 527 Patients From the Polish Adult Leukemia Group Registry. Clin Lymphoma Myeloma Leuk. 2018 Jul;18(7):e283-e285. doi: 10.1016/j.clml.2018.05.001. Epub 2018 May 9. No abstract available. PMID 29778693
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/29778693/